CLINICAL TRIAL: NCT00005833
Title: A Phase II Trial of R115777 (NSC #702818) in Patients With Advanced Colorectal Cancer
Brief Title: S9923 R115777 in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067847; S9923 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2004-04-12 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R115777 (Experimental): R115777, 300mg PO BID on Days 1-21. 1 cycle=28 days.
  Interventions: Drug: R115777

INTERVENTIONS:
Drug: R115777 — 300mg P.O. BID.
  Other Names: NSC-702818

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of R115777 in treating patients who have recurrent or advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate to R115777 in patients with disseminated colorectal cancer who have been previously treated for advanced disease. II. Assess the time to treatment failure and survival of these patients with this treatment regimen. III. Determine the frequency and severity of toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive oral R115777 twice daily on days 1-21. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study over 5-7 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced colorectal adenocarcinoma Well differentiated OR Moderately well differentiated OR Poorly differentiated Distant metastases not surgically curable Measurable disease No prior treatment for disseminated disease No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-1 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT or SGPT no greater than 2.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception Must be able to swallow or receive enteral medications through gastrostomy feeding tube No intractable nausea or vomiting No other prior malignancy for the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior adjuvant immunotherapy and recovered No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior adjuvant chemotherapy and recovered No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No more than 25% of total area of bone marrow irradiated No concurrent radiotherapy Surgery: At least 2 weeks since prior surgery and recovered Other: No concurrent proton pump inhibitors No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2000-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Confirmed complete and partial response rate to R115777 | Once every 8 weeks until progression
  Confirmed complete and partial response rate to R115777 in pts with measurable, disseminated colorectal cancer and no prior therapy for advanced disease.

SECONDARY OUTCOMES:
Time to treatment failure and survival | Once every 8 weeks until progression, then once every 6 months for 2 years, then annually until 3 years from registration
  To assess time to treatment failure and survival in this group of patients.
Frequency & severity of toxicities | Weekly for 8 weeks and then once every 4 weeks until progression
  To assess the frequency and severity of toxicities associated with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Whitehead, MD, Study Chair — University of Texas
Locations (12):
- United States (12):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Whitehead RP, McCoy S, Macdonald JS, Rivkin SE, Neubauer MA, Dakhil SR, Lenz HJ, Tanaka MS, Abbruzzese JL; Southwest Oncology Group. Phase II trial of R115777 (NSC #70818) in patients with advanced colorectal cancer: a Southwest Oncology Group study. Invest New Drugs. 2006 Jul;24(4):335-41. doi: 10.1007/s10637-005-4345-3. PMID 16683076